CLINICAL TRIAL: NCT05871710
Title: Validity and Reliability of the Turkish Version of the Tele-Pulmonary Rehabilitation Acceptance Scale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: TelePulm
Record Dates: First submitted 2023-04-27; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Disease; Telehealth; Pulmonary Rehabilitation
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in need of pulmonary rehabilitation or already receiving pulmonary rehabilitation.: Native Turkish-speaking patients in need of pulmonary rehabilitation or already receiving pulmonary rehabilitation.
  Interventions: Other: Turkish version of the Tele-Pulmonary Rehabilitation Acceptance Scale; Other: Scale Evaluation Form
- Health personnel working in the field of pulmonary rehabilitation.: Native Turkish-speaking health personnel working in the field of pulmonary rehabilitation.
  Interventions: Other: Turkish version of the Tele-Pulmonary Rehabilitation Acceptance Scale; Other: Scale Evaluation Form

INTERVENTIONS:
Other: Turkish version of the Tele-Pulmonary Rehabilitation Acceptance Scale — The Tele-Pulmonary Rehabilitation Acceptance Scale is a measuring tool that assesses the level of acceptance towards telerehabilitation programs among healthcare providers and patients in the field of pulmonary rehabilitation. It is used to evaluate the attitudes, beliefs, and perceptions of potential users towards telerehabilitation, which is a form of healthcare delivery that utilizes telecommunication technology to provide remote rehabilitation services to patients. The scale is intended to provide a standardized data collection tool that can be used to measure the level of acceptance of telerehabilitation programs among different groups of potential users. This scale will be translated into Turkish by a researcher who has an advanced level of knowledge in English and whose native language is Turkish.
Other: Scale Evaluation Form — The healthcare providers and the patients will be asked about their opinions on the scale's construction, usefulness, and scope using a 100 mm visual analog scale.

SUMMARY:
The objective of this research is to translate the Tele-Pulmonary Rehabilitation Acceptance Scale into Turkish and assess its reliability and accuracy.

DETAILED DESCRIPTION:
The use of telehealth in pulmonary rehabilitation, also known as telerehabilitation, is a novel approach in healthcare practice. In order to effectively implement telerehabilitation programs, it is important to evaluate how potential users perceive and accept this new type of program. Thus, the aim of this research was to create a measuring tool that could assess the level of acceptance of telerehabilitation among healthcare providers and patients. A group of experts in pulmonary rehabilitation, telehealth, information technology, and scale development have reviewed and confirmed the content validity of the Tele-Pulmonary Rehabilitation Acceptance Scale. This scale is significant because it offers a consistent means of collecting data to measure the level of acceptance towards telerehabilitation among potential users. This study aims to translate and show the consistency and validity of the Tele-Pulmonary Rehabilitation Acceptance Scale in Turkish.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient in need of pulmonary rehabilitation or a healthcare professional working in the field of pulmonary rehabilitation.
* Being a native Turkish speaker.
* Giving consent to participate in the study.

Exclusion Criteria:

* Any disease or condition that prevents reading, understanding, or filling out forms.
* Not giving consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Native Turkish-speaking patients in need of pulmonary rehabilitation and native Turkish-speaking healthcare professionals working in the field of pulmonary rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability of the Turkish version of the Tele-Pulmonary Rehabilitation Acceptance Scale | 1 day
  The primary outcome is the overall validity and reliability of the Turkish version of the Tele-Pulmonary Rehabilitation Acceptance Scale. This scale is a Likert scale with a total of 13 questions and the score for each question ranges from 1 to 4. The total score is 52 and higher scores indicate that the patient is more inclined to adopt telerehabilitation. This will involve analyzing the responses of participants to the questionnaire to determine if it accurately measures the intended construct. The study will also assess the internal consistency of the responses to determine if the scale produces consistent results when administered multiple times to the same group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request by the co-responding author.